CLINICAL TRIAL: NCT04289506
Title: Validation of Molecular and Protein Biomarkers in Sepsis
Acronym: VAMp-sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Public Health England (Other Government)
Collaborators: Aneurin Bevan University Health Board (Other); Cardiff University (Other)
Responsible Party: Sponsor
Other Study IDs: VAMp-Sepsis 1.1
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Sepsis; Cardiac Arrest; Pneumonia; Abdominal Sepsis; SIRS
MeSH Terms: conditions — Sepsis; Heart Arrest; Pneumonia; Intraabdominal Infections | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2.5 mL x2 blood will be collected in PAXgenes tube for mRNA extraction as well as 30mL blood for isolation of peripheral white cells (PMBC). In centres where routine clinical practice is to discard up to 5 mL blood during arterial blood gas analysis, this otherwise wasted sample will be collected in EDTA tubes for cytokine analysis (max 10 mL/day). Samples will be anonymised and processed for storage or frozen as required, within 30 minutes. Blood samples will be sent to the research consortium's approved and appointed laboratories for further analysis.
  All samples will be stored for a maximum of ten years after study closure, in order to enable validation of results with new methodology and to develop methods for detecting new biomarkers (protein and mRNA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Community-acquired pneumonia (Sepsis): Community-acquired pneumonia with organ dysfunction
  Interventions: Diagnostic Test: mRNA expression
- Abdominal sepsis: Abdominal infection due to peritoneal soiling, biliary infection, urinary tract infection leading to organ dysfunction
  Interventions: Diagnostic Test: mRNA expression
- Infection of unknown origin (Sepsis): Infection of unknown origin of less than 72 hours duration, including bacteraemia with organ dysfunction
  Interventions: Diagnostic Test: mRNA expression
- Organ dysfunction related to non-infectious cause (SIRS): Patients admitted to the ICU following out-of hospital cardiac arrest OR Patients admitted to the ICU following major trauma (ISS>12) OR Patients admitted to the ICU following pancreatitis with organ dysfunction
  Interventions: Diagnostic Test: mRNA expression
- Healthy volunteers: Healthy volunteers
  Interventions: Diagnostic Test: mRNA expression

INTERVENTIONS:
Diagnostic Test: mRNA expression — The primary objective is the external validation of our filed patent-claims panels of mRNA biomarkers, which in the inflammatory and SIRS/Sepsis panels have better discriminatory properties than any other published biomarker panel for detecting individuals with severe inflammation and differentiating infectious and non-infectious origin of organ failure (Sepsis/SIRS).

SUMMARY:
Background:

Sepsis (blood poisoning) is a clinical syndrome characterised by a dysregulated host response to infection causing life-threatening organ dysfunction which results in admission to an intensive care unit. It typically shows an initial harmful inflammation resulting from the immune system's overreaction to a severe infection. It is a major healthcare problem, affecting millions of people worldwide. In the UK, it kills over 37,000 people/year, costing the NHS £2.5 billion a year, and is increasing in incidence. Despite extensive efforts to tackle this burden, at present, however, there are no specific and effective therapies for this illness.

Sepsis is a potentially life-threatening condition caused by a severe infection. When someone develops sepsis, inflammation occurs not just at the site of the infection but throughout the whole body. This widespread inflammation can be very harmful. It is known that similar responses occur in other conditions, not relating to infection.

The investigators are recruiting patients with severe infections causing organ failure (also known as severe sepsis/ septicaemia and septic shock) and also patients where widespread inflammation, not related to infection, causes organ failure. In this study the investigators hope to find out whether certain groups of genetic and blood based protein markers of sepsis can forewarn the clinicians to this condition and also highlight patients who are responding well to the treatment.

Although it is known that the majority of the patients suffering from sepsis will survive their ICU stay and leave the hospital alive, there is insufficient data how these patients do on a longer term, i.e. after some time at home. To date there is little information on the ability of the observed genetic and blood based protein markers to predict the functional status of the patients surviving these conditions.

DETAILED DESCRIPTION:
Sepsis, defined as life threatening organ failure resulting from a dysregulated host response to infection, remains a leading cause of death in critically ill patients and has been included as a health priority in a 2017 WHO resolution. Diagnosis of this disorder is challenging because the clinical signs and symptoms of systemic inflammation in sepsis overlap with those of non-infectious critical conditions i.e. severe inflammatory response syndrome (SIRS) e.g. cardiac arrest and burns. Early and accurate diagnosis of sepsis is critical for improving patient outcomes and reducing antibiotic usage. Delays in antibiotic administration are associated with worse outcomes; however paradoxically, indiscriminate prescription of antibiotics to patients without bacterial infections increases both rates of morbidity and antimicrobial resistance. The rate of inappropriate antibiotic prescriptions in the hospital setting is estimated at 30 to 50% and would be decreased by access to improved diagnostic tests.

There is currently no gold standard laboratory test that can broadly determine the presence and type of infection. Although new polymerase chain reaction (PCR)-based molecular diagnostics can profile pathogens directly from blood culture, they suffer from sensitivity issues due to dependence on sufficient numbers of pathogens in the blood sample. They are also limited to detection of a discrete range of pathogens. As a result, there is a growing focus on molecular diagnostics that profile the host immune response. Current sepsis groupings are based on clinical criteria such as the presence of shock, infection source, or organ failure, but such groupings may not represent the underlying biology driving the host response. They have also failed to adequately match patients for novel interventions. If the heterogeneity of sepsis truly reflects heterogeneity in the host response, characterisation of these underlying host response types will be fundamental to enabling precision sepsis therapeutics.

In a previous multi-centre, clinical-temporal study in three cohorts of patients admitted to the intensive clinical care unit (ICU); (i) out of hospital cardiac arrest (n=36 - SIRS group)) (ii) pulmonary sepsis (n=84) (iii) abdominal sepsis (n=64) and 30 healthy controls, validated potential host immune biomarkers. Using 202 samples from these cohorts, the investigators derived a set of gene biomarkers which can identify patients with severe inflammation and discriminate sepsis from non-infected inflammation across a broad range of clinical conditions. Other biomarkers have been identified for use for other purposes e.g. prognosis/severity. Our patent arising from this work has been filed and entered PCT stage. From these patented markers a parsimonious set of 17 genes has been further delineated, which are under further evaluation. A sub-panel of two gene entities has been identified that can accurately detect severe inflammation using receiver operating characteristic/area under the curve (ROC) analysis with a value of approximately 0.98. A panel of three/four gene entities has been identified for discrimination of SIRS from all sepsis types (ROC 0.89-0.92), all depending on sensitivity or specificity range settings.

Better diagnostics for sepsis-driven inflammation are needed in both inpatient and outpatient settings. In low-acuity outpatient settings, contributing circa 80% of total UK antibiotic use, a simple diagnostic to discriminate a septic inflammatory process from an innocuous, self-limiting condition, would assist in appropriate antimicrobial use, appropriate triage, avoiding further investigations, and appropriate escalation / admissions. In higher-acuity settings, causes of non-infectious inflammation are important to exclude; a decision model for antibiotic prescription should include a non-infected, non-healthy cause. A reliable diagnostic, such as ours, needs to distinguish all three presentations: non-infected inflammation, sepsis, and relative health. It will represent a major step-change in provision of diagnostic/stratification capability, vastly improve decision and patient management pathways and potentially reducing antibiotic overuse in the acute medical and critical-care environment.

These biomarkers once validated in an independent cohort via qPCR for mRNA and their commensurate proteins, together with an accompanied easy-to-use, clinically oriented scoring system will represent a complete data package which can be rolled out internally, subject to the appropriate further accreditation and/or leveraged for development of point-of-care devices by commercial partners. This latter option could prove useful for dissemination of the test to other patent-appropriate global territories.

There is an urgent need to validate these findings in several ways; Using an independent patient cohort, where laboratory scientists are blinded to the clinical phenotypes of the recruited patients and clinicians are not aware of the gene expression data.

Using a bioinformatics approach to validate the results in already published datasets

This project will use different approaches to validate these novel SIRS or sepsis-associated biomarkers identified by Artificial Neural Network (ANN) and parametric data mining of previously published datasets and further validated previously from a previous well characterised clinical cohort;

1. Public Health England laboratories will assess biomarker mRNA expression using a qPCR approach, with RNA purified from patient and control whole blood
2. Public Health England and Cardiff laboratories will assess protein biomarkers using ELISA assays
3. Proteomic analysis of blood by external collaborators

Further data analysis will be conducted using ROC curve analysis and arithmetic algorithms and/or other statistical/bioinformatics methods. Assessment of specificity and sensitivity and positive and negative predictive values using well established methods will also be conducted to evaluate the performance of the biomarker panels in discriminating patient control and disease groups.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for community-acquired Sepsis and Septic Shock

  1. Age => 18
  2. Admission to hospital within 72 hours of symptoms onset and development of clinical signs of sepsis
  3. Diagnosis of sepsis

     * SEPSIS is defined as a (1) DEFINED FOCUS OF INFECTION AND (2) SOFA>2, with at least ONE organ specific SOFA subscore =2.

       1. (1) DEFINED FOCUS OF INFECTION is indicated by either i. An organism grown in blood or sterile site OR ii. An abscess or infected tissue (e.g. pneumonia, peritonitis, urinary tract, vascular line infection, soft tissue, etc).
       2. (2) The SOFA score criteria are described in the Appendix [7]
     * SEPTIC SHOCK is defined as SEPSIS plus the presence of hypotension requiring the use of vasopressors to maintain mean arterial pressure of 65 mmHg or greater and having a serum lactate level greater than 2 mmol/L persisting after adequate fluid resuscitation [8]

Inclusion Criteria for Critically Ill patients without infection

1. Patients admitted to the ICU following out-of hospital cardiac arrest OR Patients admitted to the ICU following major trauma (ISS>12) OR Patients admitted to the ICU following pancreatitis
2. Have multiorgan failure as defined by SOFA>2, with at least ONE organ specific SOFA subscore =2.
3. Patients must not be receiving antibiotics for treatment of known or suspected infection
4. patient already has or will require arterial cannulation as part of standard treatment

Exclusion Criteria:

* 1. Patients who are on immune-modulating therapy (e.g., methotrexate, prednisolone >5mg/day, or other immunosuppressants) for any length of time within 6 months of index admission 2. Patients with acquired cellular immune deficiency (E.g. active HIV infection or AIDS); 3. Patients with concurrent blood-borne viral infections (E.g. Hepatitis B or C) 4. Patients with any haematological malignancy in their past medical history; 5. Patients who are on chronic haemodialysis; 6. Solid organ transplant recipients; 7. Patients who have biopsy, image or endoscopy proven liver cirrhosis; 8. Patients who are not expected to survive beyond 90 days due to the advancement of their underlying disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with organ dysfunction due to infection and no-infectious causes.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
mRNA expression levels | Day 1 ICU/Hospital admission
  mRNA expression levels from peripheral blood cells

SECONDARY OUTCOMES:
Mortality | 30 days
  All-cause mortality
Mortality | 90 days
  All-cause mortality
Health related quality of life | 6 months
  EuroQol Group 5 Domain questionnaire (EQ-5D). Range 1 to 5 in the domains. Higher values indicate worse health outcomes in the subdomains.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Aneurin Bevan University Health Board, Newport, Gwent
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Public Health England, London

IPD SHARING:
Plan to Share IPD: No
Requests for access to study data will be considered, and approved in writing where appropriate, after formal application to the Chief Investigator.

REFERENCES:
- [Background] Reinhart K, Daniels R, Kissoon N, Machado FR, Schachter RD, Finfer S. Recognizing Sepsis as a Global Health Priority - A WHO Resolution. N Engl J Med. 2017 Aug 3;377(5):414-417. doi: 10.1056/NEJMp1707170. Epub 2017 Jun 28. No abstract available. PMID 28658587
- [Background] Cohen J, Vincent JL, Adhikari NK, Machado FR, Angus DC, Calandra T, Jaton K, Giulieri S, Delaloye J, Opal S, Tracey K, van der Poll T, Pelfrene E. Sepsis: a roadmap for future research. Lancet Infect Dis. 2015 May;15(5):581-614. doi: 10.1016/S1473-3099(15)70112-X. Epub 2015 Apr 19. PMID 25932591
- [Background] Sweeney TE, Shidham A, Wong HR, Khatri P. A comprehensive time-course-based multicohort analysis of sepsis and sterile inflammation reveals a robust diagnostic gene set. Sci Transl Med. 2015 May 13;7(287):287ra71. doi: 10.1126/scitranslmed.aaa5993. PMID 25972003
- [Background] Sweeney TE, Thomas NJ, Howrylak JA, Wong HR, Rogers AJ, Khatri P. Multicohort Analysis of Whole-Blood Gene Expression Data Does Not Form a Robust Diagnostic for Acute Respiratory Distress Syndrome. Crit Care Med. 2018 Feb;46(2):244-251. doi: 10.1097/CCM.0000000000002839. PMID 29337789
- [Background] Kempsell KE, Ball G, Szakmany T. Issues in biomarker identification, validation and development for disease diagnostics in Public Health. Expert Rev Mol Diagn. 2016;16(4):383-6. doi: 10.1586/14737159.2016.1133300. Epub 2016 Jan 22. No abstract available. PMID 26680111
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- See also: Patent description of mRNA marker sets validated — https://patents.google.com/patent/WO2018060739A2/